CLINICAL TRIAL: NCT05810571
Title: Comparison of Erector Spina and Quadratus Lumborum in Open Nephrectomy
Brief Title: Comparison of Postoperative Analgesic Efficacy of the Erector Spina Plane Block and Quadratus Lumborum Block in Open Nephrectomy: a Prospective Randomized Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: KAEK / 12bl.01
Record Dates: First submitted 2023-03-31; First posted 2023-04-12 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-09

CONDITIONS: Renal Cell Carcinoma
Keywords: erector spina plane block; quadratus lumborum block; patient controlled analgesia; nephrectomy; analgesia
MeSH Terms: conditions — Carcinoma, Renal Cell; Agnosia | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: participant will not know which block applied, and the outcome assessor of the postoperative analgesia will not know
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- patient controlled analgesia (Placebo Comparator): this group of patients received no block, received only postoperative patient-controlled analgesia with morphine
  Interventions: Procedure: preoperative remifentanil consumption; Procedure: postopeartive controlled anlagesia with morphine
- erector spina plane block (Active Comparator): this group of patients received erector spina plane block preoperatively, received only postoperative patient-controlled analgesia with morphine
  Interventions: Procedure: preoperative remifentanil consumption; Procedure: postopeartive controlled anlagesia with morphine
- quadratus lumborum block (Active Comparator): this group of patients received erector spina plane block preoperatively, received only postoperative patient-controlled analgesia with morphine
  Interventions: Procedure: preoperative remifentanil consumption; Procedure: postopeartive controlled anlagesia with morphine

INTERVENTIONS:
Procedure: preoperative remifentanil consumption — continuous remifentanil infusion will applied for peroperative analgesia
Procedure: postopeartive controlled anlagesia with morphine — postoperative morphine patient controlled analgesia will be applied for postoperative analgesia

SUMMARY:
patients who will undergo elective open nephrectomy will be divided into three groups; the control (PCA), the erector spina plane block, and the quadratus lumborum block. After standard anesthesia induction and monitorization then Bispectral index monitoring will be applied to all patients. Anesthesia will be maintained using sevoflurane in a mixture of oxygen and air. Continuous remifentanil infusion will be used for analgesia. Then patient's numeric rating scales and morphine pca consumptions will be recorded for one day.

DETAILED DESCRIPTION:
patients who will undergo elective open nephrectomy will be divided into three groups; the control (PCA), the erector spina plane block and the quadratus lumborum block. After standard anesthesia induction and monitorization then Bispectral index monitoring will be applied to all patients. Anesthesia will be maintained using sevoflurane in a mixture of oxygen and air. Continious remifentanil infusion will be used for analgesia. Then patient's numeric rating scales and morphine pca consumptions will be recorded for one day.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* open nephrectomy elective patients
* BMI<35

Exclusion Criteria:

* ASA 4-5-6
* Laparoscopic nephrectomy
* infection at the block side
* coagulation disorder
* BMI>35

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2027-01-03 (Estimated); Study Completion 2027-01-03 (Estimated)

PRIMARY OUTCOMES:
postoperative morphine consumption | 24 hour postoperatively
  amount of postoperative morphine use of the patient's

SECONDARY OUTCOMES:
peroperative remifentanil consumptions | 4 hour preoperatively
  amount of remifentanil use of the patient's
numeric rating scale | 24 hour postoperatively
  numeric rating scores of the patient's postoepartively

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Kocaeli University Medical Faculty, İzmit
  - Kocaeli University Medical Faculty, Kocaeli

IPD SHARING:
Plan to Share IPD: No